CLINICAL TRIAL: NCT02879487
Title: Vaginal Cuff Dehiscence After Two Different Colpotomy Techniques at Total Laparoscopic Hysterectomy; a Randomized Clinical Trial
Brief Title: Vaginal Cuff Dehiscence at Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, salih taskin, Assoc Prof, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2016-08-19; First posted 2016-08-25 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Surgical Wound Dehiscence
MeSH Terms: conditions — Surgical Wound Dehiscence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coagulation mode (Active Comparator): Colpotomy will be performed by monopolar needle electrode using coagulation mode
  Interventions: Device: Monopolar needle electrode
- Cut mode (Active Comparator): Colpotomy will be performed by monopolar needle electrode using cut mode
  Interventions: Device: Monopolar needle electrode

INTERVENTIONS:
Device: Monopolar needle electrode — Colpotomy during total laparoscopic hysterectomy

SUMMARY:
The aim of this study is to assess a major complication of total laparoscopic hysterectomy, vaginal dehiscence, with two different colpotomy techniques. With this aim patients to be operated for laparoscopic hysterectomy will be randomized to two different techniques. The colpotomy will be undertaken by 'cut mode' in the first group and 'coagulation mode' in the second group. All of the operations will be preformed by the same surgical at a university hospital. Vaginal dehiscence after surgery is the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* All total laparoscopic hysterectomies performed by a single surgeon
* Both benign and malignant cases
* Completed laparoscopically
* Intracorporeal vaginal cuff suturing

Exclusion Criteria:

* Robotic hysterectomies
* Pelvic infection within 30 days before surgery
* Conversion to laparotomy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-08; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Vaginal dehiscence | 3 months
  Vaginal dehiscence up to 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Emre Şükür, MD, Study Chair — Ankara University
Locations (1):
- Ankara University Medical Faculty Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes